CLINICAL TRIAL: NCT00704093
Title: The Effect of Right Ventricular Pacing on Myocardial Oxidative Metabolism and Efficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Juhani Knuuti, Director, Turku PET Centre
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 2442007§149
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-07

CONDITIONS: Bradycardia
Keywords: pacing; perfusion; oxidative metabolism; efficiency
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Right ventricular pacing — Right ventricular pacing vs. sinus rhythm or atrial pacing at the same rate

SUMMARY:
Right ventricular (RV) apical pacing induces a left bundle branch block (LBBB) type electrical activation sequence in the heart. This abnormal activation pattern of the ventricles may have detrimental effects on cardiac structure and function. RV pacing has been shown to impair left ventricular (LV) function both in normal and failing hearts. Importantly, it has been demonstrated that this deterioration in LV function is related to the presence of LV dyssynchrony during RV pacing.

The exact effects of RV pacing on myocardial perfusion, oxidative metabolism and cardiac efficiency have not been fully elucidated. The objective of the present study is to evaluate the effect of RV pacing on both global and regional oxidative metabolism and perfusion, and myocardial efficiency. In addition, the effect of RV pacing induced LV dyssynchrony on myocardial oxidative metabolism and efficiency will be studied.

Our hypothesis is that LV dyssynchrony during RV pacing results in regional abnormalities in LV perfusion and oxidative metabolism. LV dyssynchrony will also result in altered myocardial efficiency.

DETAILED DESCRIPTION:
Right ventricular (RV) apical pacing induces a left bundle branch block (LBBB) type electrical activation sequence in the heart. This abnormal activation pattern of the ventricles may have detrimental effects on cardiac structure and function. Several clinical trials have demonstrated an association between RV pacing and an increased risk of heart failure and death. In addition, RV pacing has been shown to impair left ventricular (LV) function both in normal and failing hearts. Importantly, it has been demonstrated that this deterioration in LV function is related to the presence of LV dyssynchrony during RV pacing.

The exact effects of RV pacing on myocardial perfusion, oxidative metabolism and cardiac efficiency have not been fully elucidated. Importantly, the relation between the presence of LV dyssynchrony during RV pacing and changes in myocardial perfusion, oxidative metabolism and cardiac efficiency has not been studied.

Ten patients with normal LV ejection fraction and VVI/DDD pacemaker will be studied during AAI-pacing/sinus rhythm without RV pacing (pacing-OFF) and with RV-pacing (pacing-ON) at the same heart rate. Dynamic [15O]water and [11C]acetate positron emission tomography is used to measure perfusion and oxidative metabolism (kmono) of the LV. An echocardiographic examination is used to assess LV stroke volume (SV) and LV dyssynchrony.

The PET data will be first analyzed based on RV pacing mode only, comparing the two pacing conditions (pacing-ON vs. pacing-OFF). Thereafter, the study population will be divided into two groups, according to the presence of LV dyssynchrony during RV pacing.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age over 18 years
* Previously implanted permanent pacemaker (DDD or VVI)
* Normal left ventricular function

Exclusion Criteria:

* Pacemaker dependency
* Symptomatic coronary artery disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
myocardial perfusion, oxidative metabolism and efficiency | At baseline and at 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Juhani Knuuti, MD, prof, Study Director — Turku PET Centre
Locations (1):
- Turku PET Centre, Turku, Finland